CLINICAL TRIAL: NCT06313307
Title: The Efficacy in Treatment of Facial Melasma Combined With Thulium 1927-nm Fractional Laser and Topical H2R Antagonist: a Split-face, Single-blind Study
Brief Title: The Efficacy in Treatment of Facial Melasma Combined With Thulium 1927-nm Fractional Laser and Topical H2R Antagonist
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: famotidine and melasma
Record Dates: First submitted 2024-02-29; First posted 2024-03-15 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: Melasma
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thulium 1927nm fractional laser (Active Comparator): 1927nm fractional laser (South Korea, WONTECH, Lavieen) was performed with 4-week interval (Week 0, 4, 8, 12 and 16) for a total of 4 treatments. The parameter of 1927nm fractional laser was as follows: duration 600-800um, 10w, density 0.8mm, 1 pass.
  Interventions: Device: Thulium 1927-nm Fractional Laser
- Thulium 1927nm fractional laser and topical H2R antagonist (Experimental): Topical H2RA (2% famotidine solution solved in double-distilled water (containing poloxamer 407, glycerol, lauryl alcohol polyether-4, polyethylene glycol-8, and propylene glycol)) was applied immediately after the laser therapy and then topically twice per day in the morning and the evening for 16 weeks.
  Interventions: Combination Product: topical H2R antagonist; Device: Thulium 1927-nm Fractional Laser

INTERVENTIONS:
Combination Product: topical H2R antagonist — Topical H2RA (2% famotidine solution solved in double-distilled water (containing poloxamer 407, glycerol, lauryl alcohol polyether-4, polyethylene glycol-8, and propylene glycol)) was applied topically twice per day in the morning and the evening for 16 weeks.
  Arms: Thulium 1927nm fractional laser and topical H2R antagonist
Device: Thulium 1927-nm Fractional Laser — 1927nm fractional laser (South Korea, WONTECH, Lavieen) was performed with 4-week interval (Week 0, 4, 8, 12 and 16) for a total of 4 treatments. The parameter of 1927nm fractional laser was as follows: duration 600-800um, 10w, density 0.8mm, 1 pass.

SUMMARY:
Melasma is a hyperpigmentary disorder of the skin especially of the face. Compared with normal skin, histologic features of melasma include the enhanced activity of melanocytes, higher solar elastosis in upper dermis, basement membrane disruption which promotes melanocytes and melanin into the dermis, increased vascularization, and an increased number of mast cells.

1927nm fractional laser was approved to treat melasma with no major side effects, however,hyperpigmentation and recurrence occasionally happened after laser therapy. Mast cells may paly a key role in the refractory melasma and hyperpigmentation. We hypothesized that laser treatment may stimulate the activation of pre-existing mast cell in melasma skin and promote mast cell proliferation and degranulation to release mediators such as histamine (HA). HA has been demonstrated to increase the melanin content and tyrosinase activity of melanocytes and induce melanogenesis and morphological changes by activating cAMP-PKA pathway through H2 receptors on melanocytes5. H2R antagonist(H2RA) can suppress pigmentation by reducing the increase of activated melanocytes by UVB irradiation.

In the present study, the investigators speculated that H2RA can enhance the efficacy of laser treatment of melasma and block the histamine-mediated melanogenesis and dendricity to prevent postoperative hyperpigmentation. The investigators combined 1927nm fractional laser with topical famotidine for melasma as a new therapeutic strategy to treat melasma.The investigators performed a split-face, single-blinded study to evaluate the efficacy and safety of 1927nm fractional laser with topical famotidine for the treatment of facial melasma.

DETAILED DESCRIPTION:
Melasma is a common hyperpigmented skin disorder presented with light to dark symmetrical brown macules on face, malar and forehead areas in women with Fitzpatrick type III-IV. Compared with normal skin, histologic features of melasma include the enhanced activity of melanocytes, higher solar elastosis in upper dermis, basement membrane disruption which promotes melanocytes and melanin into the dermis, increased vascularization, and an increased number of mast cells1. As a result, melasma is often difficult to treat and is prone to recurrence.

The pathophysiology of melasma is complex and has not been fully elucidated. Possible pathogenesis of melasma includes ultraviolet (UV) exposure, genetic factors, sex hormones2, chronic skin inflammation, skin barrier disfunction also contributes in the onset of melasma1. Albeit melasma represents as melanin overproduction, multiple cell types are implicated in the pathogenesis of melasma.

Mast cell number is increased in the dermis of melasma skin, especially in the areas with solar elastosis3. Studies shown that the number of mast cells may be related to refractory and recurrence of melasma treatment4. Though the role of mast cells in the development of melasma remains unclear, based on the previous studies, among the bioactive mediators released by mast cells, histamine plays a pivotal role in UV-induced activation of melanocytes5. There are 4 subtypes of histamine receptors (HR1-4)6. Among the 4 subtypes of HRs, histamine stimulates melanocyte activation through H2 receptors on melanocytes7.The function of H2R activation has been verified in vivo by a UV-induced pigmentation in guinea pig5. Some therapeutic drugs for melasma such as tranexamic acid, corticosteroids and calcineurin inhibitors can inhibit the recruitment and maturation of mast cell by inhibiting mast cell proliferation3. These drugs inhibit melanocyte activation by reducing inflammation in melasma skin, while H2 receptor antagonists (H2RA) suppress pigmentation by inhibiting histamine-mediated melanogenesis and dendricity rather than preventing the inflammation induction. Thus, H2- blockers such as famotidine as a potential treatment strategy for melasma should be valued. The latest clinical trials have shown possible benefits of the oral H2-blocker famotidine combined with H1-blocker ketotifen for melasma8. This report provides more evidence for the efficacy of H2RA famotidine in melasma. However, the function of famotidine should be evaluated. Moreover, topical administration of famotidine may offer greater benefits than oral medication, but the effect should be evaluated further.

Lasers and light-based devices such as low-fluence Q-switched 1064-nm Nd:YAG laser have been considered as an effective modality for the treatment of melasma by directly targeting melanosome9,10. The non-ablative 1927 nm fractional thulium fiber laser targets water instead of melanocytes and conferring greater ability to target superficial layers of the skin11, thus has less risk of PIH than melanosome targeting lasers. Also, the fractional laser induced microscopic treatment zones (MTZs) can promote local drug absorption and bioavailability while reducing the undesirable effects associated with systemic absorption.12

In the present study, The investigators attempted to verified role of H2R inhibitor in the treatment of melasma by combining famotidine with 1927nm fractional laser-assisted drug delivery13. The investigators performed a split-face, single-blinded study to evaluate the efficacy and safety of 1927nm fractional laser with topical famotidine for the treatment of facial melasma.

ELIGIBILITY:
Inclusion Criteria:

* Patients with symmetrical melasma on both sides of the face were included

Exclusion Criteria:

* allergic to the famotidine;
* pregnant or lactating
* received other treatment for melasma in the last 1 month
* taking contraceptive pills for a long time
* with skin cancer, systemic diseases or mental illness
* patients with active inflammation or viral infection on the face
* patients with a history of facial injections or surgery in the 2 months prior to the test
* patients with immunodeficiency diseases
* patients with the need to work outdoors for long periods of time and who are unable to protect themselves from the sun.

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2023-04-01 (Actual); Primary Completion 2023-11-25 (Actual); Study Completion 2023-11-25 (Actual)

PRIMARY OUTCOMES:
Modified Melasma Area Severity Score（mMASI） | week0，4，8，12，16
  Minimum 0 points, maximum 7.2 points. The higher the score, the more severe the lesions

SECONDARY OUTCOMES:
melanin index（MI） | week0，4，8，12，16
  The melanin content of the skin,the higher the score, the more severe the lesions
erythema index(EI) | week0，4，8，12，16
  The severity of erythema of skin, the higher the score, the more severe the lesions

OTHER OUTCOMES:
Melasma Quality of Life Index(MELASQoL) | week 0 and week 16
  The higher the score, the more melasma affects the patient

CONTACTS AND LOCATIONS:
Overall Officials: ZHAO WANG, Study Director — The second affiliated hospital of Xian Jiaotong University
Locations (1):
- The second affiliated hospital of Xi'an Jiaotong University, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No